CLINICAL TRIAL: NCT05667857
Title: Longitudinal Neurocognitive, Psychosocial and Health-related Quality of Life Assessment in Advanced Cancer Survivors Treated With Immunotherapy and the Efficacy of Integrative Neurocognitive Remediation Therapy
Acronym: CognIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Bart Neyns, Prof. Dr., Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-BN-001
Record Dates: First submitted 2022-07-14; First posted 2022-12-29 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Remediation; Neuropsychology; Quality of Life; Psycho-Oncology; Cognitive Behavioral Therapy; Cancer Survivors; Immunotherapy; Cognitive Dysfunction; Psychological Distress
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: We will have three cohorts:
  * Cohort 1: advanced cancer survivors treated with immunotherapy
  * Cohort 2: cancer survivors treated with cancer therapy of any kind (excluded immunotherapy)
  * Cohort 3: cancer survivors of a CNS tumor, who do not have active disease in the CNS
  All patients of cohort 1 will receive a psychosocial and neurocognitive assessment at baseline. Patients who do not have cognitive problems or do not have interest in following the integrative neurocognitive remediation therapy program will go into the non-intervention group for follow-up.
  Patients of cohort 1, 2 and 3 who have cognitive problems and/or cognitive complaints who want to follow the integrative neurocognitive remediation program will complete a neurocognitive and psychosocial assessment before and immediately after the remediation program. The same assessment will be repeated six months after finishing the therapy program, to investigate the long-term efficacy of the therapy program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-intervention group (No Intervention): These participants will a undergo a neurocognitive and psychosocial assessment at baseline, and in follow-up after 6 months and 1 year thereafter. The aim of this group is to measure the extent of psychosocial and cognitive difficulties and health-related quality of life.
- Integrative neurocognitive remediation therapy (Experimental): The experimental group will undergo profound neuropsychological and psychological assessment before starting the integrative neurocognitive remediation therapy, in addition to the assessment already done at baseline. This group will repeat the testing after completion of the integrative neurocognitive remediation therapy, and 6 months thereafter.
  Interventions: Behavioral: Integrative neurocognitive remediation therapy

INTERVENTIONS:
Behavioral: Integrative neurocognitive remediation therapy — Integrative Neurocognitive Remediation Therapy is a clinical program of 12 weeks (1 day/week) that combines personalized computerized cognitive training and neurocognitive strategy training, with group sessions of adapted physiotherapy, acceptance and commitment therapy (ACT), cognitive behavioral therapy (CBT) and information sessions on cognition, fatigue, nutrition and physical exercise.
  Arms: Integrative neurocognitive remediation therapy

SUMMARY:
Since 2010, the field of immunotherapy has grown substantially, leading to a growing population of long-term cancer survivors treated with immunotherapy. Since cancer survivorship in immunotherapy is an emerging field, to date not much is known about psychosocial and neurocognitive survivorship-related issues in advanced cancer survivors treated with immunotherapy. Preliminary findings indicated significant psychosocial and cognitive problems in survivors of advanced melanoma persist after treatment with immunotherapy. The objective for this project is twofold. First, the investigators want to longitudinally identify survival-related problems in survivors of advanced cancer treated with immunotherapy. The second goal is to identify the efficacy of an Integrative Neuro-Cognitive Remediation Therapy (INCRT) program. The investigators will focus on the following outcomes: (1) Psychosocial consequences, such as emotional complaints, fatigue, fear of recurrence, (2) neurocognitive functioning, and (3) health-related quality of life. The INCRT combines personalized computerized cognitive training and neurocognitive strategy training, with group sessions of exercise, mindfulness, Acceptance and Commitment Therapy, and cognitive behavioral therapy.

We will have three cohorts:

* Cohort 1: advanced cancer survivors treated with immunotherapy
* Cohort 2: cancer survivors treated with cancer therapy of any kind (excluded immunotherapy), and who have subjective complaints and/or objective cognitive impairment
* Cohort 3: cancer survivors of a central nervous system (CNS) tumor, who do not have active disease in the CNS, and who have subjective complaints and/or objective cognitive impairment

In the first part of the study, survival-related problems will be evaluated in cohort 1, in a longitudinal manner by means of a semi-structured interview at baseline, various questionnaires and a computerized neuropsychological test battery.

In the second part of the study, patients of cohort 1, 2 and 3 with subjective or objective cognitive dysfunction can follow the INCRT program. The efficacy of the INCRT is evaluated through a pre-INCRT and post-INCRT evaluation. This evaluation consist of several questionnaires and neuropsychological tests. Long-term efficacy will be evaluated by a follow-up evaluation six months after completion of the INCRT program.

ELIGIBILITY:
Inclusion Criteria:

1. Non-intervention group:

   * Provision of written informed consent
   * Diagnosed with advanced cancer of any type
   * Initiated immunotherapy (Anti-PD1, Anti-PDL1, CTLA-4, …) at least one year ago
   * Have a confirmed normalization on whole-body 18F-FDG PET
   * English, Dutch or French-speaking
2. Integrative neurocognitive remediation therapy group:

   * Provision of written informed consent
   * Objective cognitive impairment and/or subjective cognitive complaints
   * Confirmed normalization on whole-body 18F-FDG PET for patients (cohort 1)
   * Disease-free (cohort 2) or no active disease for patients with CNS tumors (cohort 3)
   * Having received a cancer therapy of any kind
   * Having ended cancer treatment (immunotherapy, chemotherapy, radiotherapy, surgery, …) with an exception of ongoing adjuvant hormone therapy
   * Dutch or French speaking

Exclusion Criteria:

* severe co-morbid non cancer-related psychiatric disorders such as psychosis, obsessive compulsive disorders, eating disorders etc., patients with cognitive impairment related to dementia, and patients that are physically or mentally not able to fill in the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Objective neurocognitive functioning measured by the COGBAT neuropsychological battery. | Until study completion, with an average of 3 years
  To measure neurocognitive functioning (attention, memory and executive functioning), with the computerized neuropsychological test battery COGBAT. This battery gives an overall degree of objective neurocognitive functioning, in addition to the specific test performance per subtest. The test performance will be measured in raw scores and z-scores. This test battery will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. Improvement in test performance after the therapy program, compared to baseline, will indicate efficacy of the integrative neurocognitive remediation therapy program.
Subjective cognitive complaints measured by the Cognitive Failures Questionnaire. | Until study completion, with an average of 3 years
  To measure subjective cognitive functioning as assessed by the Cognitive Failures Questionnaire, values ranging from 0 to 100. Higher values mean more cognitive complaints. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. A cut-off score of 44 will be used to define elevated levels of cognitive complaints, a score higher than 54 indicates severe cognitive complaints. Improvement in subjective cognitive complaints after the therapy program, compared to baseline, will indicate efficacy of the integrative neurocognitive remediation therapy program.
Emotional distress as assessed by the Hospital Anxiety and Depression Scale. | Until study completion, with an average of 3 years
  To identify emotional distress, the Hospital Anxiety and Depression Scale will be used, with values ranging from 0 to 42. Higher scores mean more emotional distress. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. A cut-off score of 8 will be used to define elevated levels of emotional distress, a score higher than 10 corresponds to moderate emotional distress, a score higher than 14 corresponds to severe emotional distress.
Fatigue as assessed by Fatigue Severity Scale. | Until study completion, with an average of 3 years
  To identify fatigue, the Fatigue Severity Scale will be used. Mean scores will be calculated, leading to a score between 1 and 7. Higher values indicate more fatigue. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. A cut-off score of 4 will be used to define elevated levels of fatigue.
Fear of cancer recurrence as assessed by the Fear of Cancer Recurrence Inventory-Short Form (FCRI-SF). | Until study completion, with an average of 3 years
  To identify fear of cancer recurrence, the Fear of Cancer Recurrence Inventory-Short Form (FCRI-SF). will be used. Values range from 0 to 36 and higher values indicate more fear of cancer recurrence. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. A cut-off score of 13 will be used to define significant fear of cancer recurrence. A score higher than 15 equals clinically significant fear of cancer recurrence, a score higher than 21 equals a pathological fear of cancer recurrence.
Health-related quality of life as assessed by the EORTC Quality of Life Core 30 Questionnaire. | Until study completion, with an average of 3 years
  To measure health-related quality of life, the EORTC Quality of Life Questionnaire (EORTC-QLQ-C30) will be used. Transformed scores range between 0 and 100, higher scores indicate better health-related quality of life. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. The scores will be compared to the Threshold of Clinical Importance, developed by Giesinger et al. (2020). To evaluate change over time, the changes of at least 10 points are regarded, which are supported to be clinically meaningful changes (Snyder et al., 2014).

SECONDARY OUTCOMES:
To document baseline demographic data, prior disease history, nature of immunotherapy therapy | Baseline
  To document baseline demographic data, prior disease history, nature of immunotherapy therapy, the investigators will look into the patient medical record and a general questionnaire will be used.
To measure the feasibility of the implementation in a larger scale of this clinical cognitive rehabilitation program for cancer survivors, as assessed by the resources needed to implement this program. | Until study completion, with an average of 3 years
  To explore the feasibility of the implementation in a larger scale of this clinical program will be assessed by the care need of the patients and the possibility to implement the therapy program in other hospitals (resources needed, cost of the program for the patient).
To measure the relation between psychological distress, as assessed by the Hospital Anxiety and Depression Scale, and subjective cognitive functioning, as assessed by the Cognitive Failures Questionnaire. | Until study completion, with an average of 3 years
  Psychological distress will be measured by the sum scores of the Hospital Anxiety and Depression Scale. Subjective cognitive functioning will be measured by the sum scores of the Cognitive Failures Questionnaire. To measure the relation between the two variables, the investigators will conduct a statistical correlation of these outcomes. The outcome will be a correlation coefficient (r).
To measure the relation between psychological distress, as assessed by the Hospital Anxiety and Depression Scale, and objective cognitive functioning, as assessed by the COGBAT neuropsychological battery. | Until study completion, with an average of 3 years
  Psychological distress will be measured by the sum scores of the Hospital Anxiety and Depression Scale. Objective cognitive functioning will be measured by the COGBAT neuropsychological battery. To measure the relation between the two variables, the investigators will conduct a statistical correlation of these outcomes. The outcome will be a correlation coefficient (r).
To measure the relation between subjective neurocognitive functioning, as assessed by the Cognitive Failures Questionnaire, and the objective cognitive functioning, as assessed by the COGBAT neuropsychological battery. | Until study completion, with an average of 3 years
  Subjective cognitive functioning will be measured by the sum scores of the Cognitive Failures Questionnaire. Objective cognitive functioning will be measured by the COGBAT neuropsychological battery. To measure this relation, the investigators will conduct a statistical correlation of these outcomes. The outcome will be a correlation coefficient (r).
To explore the care needs of personalized nutritional advice. | Until study completion, with an average of 3 years
  This will be assessed through two open questions asked to the patient, more specifically: 1) if the patient has interest in personalized nutritional advice, 2) what the specific nutritional care need is of the patient.
Rumination as assessed by the Brooding items of the Ruminative Response Scale (RRS). | Until study completion, with an average of 3 years
  To identify rumination, the Brooding items of the Ruminative Response Scale (RRS) will be used. Values range from 5 to 20, higher values indicate more tendency of 'Brooding', a maladaptive type of rumination. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter.
Visuo-spatial short-term memory measured by the computerized version of the Corsi Block Tapping Test by the Vienna Test System | Until study completion, with an average of 3 years
  To measure visuo-spatial memory span, with the computerized version of the Corsi Block Tapping Test by the Vienna Test System. The test performance will be measured in raw scores and z-scores. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter.
Verbal long-term memory measured by the California Verbal Learning Test | Until study completion, with an average of 3 years
  To measure verbal long-term memory measured by the California Verbal Learning Test. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and six months thereafter. The test performance will be measured in raw scores and z-scores.
Information processing speed measured by the WAIS-IV Symbol Search and Coding | Until study completion, with an average of 3 years
  To measure information processing speed measured by the WAIS-IV Symbol Search and Coding. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and six months thereafter. The test performance will be measured in raw scores and Weschler subscale scores. The Weschler subscale scores range from 0-20 and have a mean of 10.
Verbal short-term memory measured by the WAIS-IV Digit Span Forwards | Until study completion, with an average of 3 years
  To measure verbal short-term memory by the WAIS-IV Digit Span Forwards. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and six months thereafter. The test performance will be measured in raw scores and z-scores.
Working memory measured by the WAIS-IV Digit Span Backwards | Until study completion, with an average of 3 years
  To measure working memory by the WAIS-IV Digit Span Backwards. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and six months thereafter. The test performance will be measured in raw scores and z-scores.
Anxiety as assessed by the State-Trait Anxiety Inventory | Until study completion, with an average of 3 years
  Anxiety will be measured by the State-Trait Anxiety Inventory. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and 6 months thereafter. Values range from 20 to 80. Higher values indicate more anxiety. STAI scores classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Self-esteem as assessed by the Rosenberg Self-Esteem Scale. | Until study completion, with an average of 3 years
  Self-esteem will be measured by the Rosenberg Self-Esteem Scale. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and 6 months thereafter. Values range from 0 to 30. Higher values indicate a higher self-esteem. Scores between 15 and 25 are within normal range; scores below 15 correspond to low self-esteem.
Tendency for procrastination as assessed by the Pure Procrastination Scale. | Until study completion, with an average of 3 years
  Tendency for procrastination will be measured by the Pure Procrastination Scale. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and six months thereafter. Values range from 11 to 55. Higher values indicate more tendency for procrastination. A score lower than 28 indicate a low level of procrastination, a score between 28-39 indicate a moderate level of procrastination, and a score higher than 39 indicate a high level of procrastination.
Metacognition as assessed by the Metacognition Questionnaire. | Until study completion, with an average of 3 years
  Metacognition will be measured by the Metacognition Questionnaire. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and six months thereafter. Values range from 30 to 120. Higher values indicate more metacognitive beliefs.
Tendency for perfectionism as assessed by the Frost Multidimensional Perfectionism Scale. | Until study completion, with an average of 3 years
  Tendency for perfectionism will be measured by the Frost Multidimensional Perfectionism Scale. This will be tested only in the intervention group, i.e. the patients that will follow the integrative neurocognitive remediation therapy. It will be repeated after completion of the therapy program and six months thereafter. Values range from 35 to 210, higher values indicate more tendency for perfectionism.
Post-traumatic stress disorder symptoms as assessed by the PTSD checklist for DSM-5 (PCL-5). | Until study completion, with an average of 3 years
  To identify post-traumatic stress disorder (PTSD) symptoms, the PTSD checklist for DSM-5 (PCL-5) will be used. Values range from 0 to 80, and higher values indicate more symptoms of post-traumatic stress. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. A cut-off score of 33 indicates PTSD.
Subjective cognitive complaints measured by the cognitive functioning subscale of the EORTC QLQ-C30. | Until study completion, with an average of 3 years
  To measure subjective cognitive functioning as assessed by the EORTC QLQ-C30, cognitive functioning subscale. Transformed scores range from 0 to 100, with higher scores meaning better cognitive functioning. This will be repeated during follow-up for the non-intervention group. For the intervention group, the scores will be compared before and after the integrative neurocognitive remediation therapy, and 6 months thereafter. The scores will be compared to the Threshold of Clinical Importance, developed by Giesinger et al. (2020). To evaluate change over time, the changes of at least 10 points are regarded, which are supported to be clinically meaningful changes (Snyder et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - University Hospital Brugmann, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel, Brussels, Brussels Capital

IPD SHARING:
Plan to Share IPD: No